CLINICAL TRIAL: NCT00469313
Title: Efficacy of Inspiratory Muscle Training on Inspiratory Capacity in Patients
Brief Title: Efficacy of Inspiratory Muscle Training on Inspiratory Capacity in Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hospital Hietzing (Other)
Other Study IDs: L1234
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: COPD
Keywords: copd; inspiratory muscle training; IF
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis:benefits of inspiratory muscle strenght training with Respifit S decreases symptoms, disability or handicap of patients affected by COPD. The inspiratory fraction (inspiratory capacity IC/ total lung capacity TLC)may be functionally more representative than other traditional indices.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD II-III (FEV1<80 and >30%)

Exclusion Criteria:

* Pregnancy
* Lung cancer
* Diabetes mellitus
* Primary exacerbation of COPD

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reiter, Study Chair — Hospital Hietzing, A 1130, Vienna, Austria
Locations (1):
- Hospital Hietzing, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Petrovic M, Reiter M, Zipko H, Pohl W, Wanke T. Effects of inspiratory muscle training on dynamic hyperinflation in patients with COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:797-805. doi: 10.2147/COPD.S23784. Epub 2012 Nov 30. PMID 23233798